CLINICAL TRIAL: NCT04394598
Title: A Phase II Randomized Study of the Protection Effect of Chinese Herbal Compound Dendrobium Huoshanense Granules in NCRT for Patients With Locally Advanced Rectal Cancer
Brief Title: A Study of Chinese Herbal Compound Dendrobium Huoshanense Granules in NCRT for Patients With Locally Advanced Rectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhu Ji, Clinical Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FDRT-R20
Record Dates: First submitted 2020-05-13; First posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Locally Advanced Rectal Cancer
Keywords: Neoadjuvant Chemoradiotherapy; Dendrobium Huoshanense; irinotecan; capecitabine
MeSH Terms: interventions — Capecitabine; Irinotecan

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRT with Dendrobium Huoshanense (Experimental): Dendrobium Huoshanense Granules: 3g tid per day for 5weeks
  Concurrent Chemoradiotherapy:
  Radiation: 50Gy/25Fx; Capecitabine: 625mg/m2 bid Monday-Friday per week; Irinotecan: 80mg/m2 (UGT1A1*28 6/6) or 65mg/m2 (UGT1A1*28 6/7)
  Chemotherapy in Interval Between CRT and Surgery:
  Capecitabine: 1000mg/m2 bid d1-14; Irinotecan: 200mg/m2 d1
  Surgery:
  Scheduled 6-8 weeks after the completion of CRT Adjuvant Chemotherapy: depends on patients pathological review.
  Interventions: Drug: Dendrobium Huoshanense Granules; Radiation: Pelvic Radiation; Drug: Capecitabine; Drug: Irinotecan
- CRT with Placebo (Placebo Comparator): Placebo: 3g tid per day for 5weeks
  Concurrent Chemoradiotherapy:
  Radiation: 50Gy/25Fx; Capecitabine: 625mg/m2 bid Monday-Friday per week; Irinotecan: 80mg/m2 (UGT1A1*28 6/6) or 65mg/m2 (UGT1A1*28 6/7)
  Chemotherapy in Interval Between CRT and Surgery:
  Capecitabine: 1000mg/m2 bid d1-14; Irinotecan: 200mg/m2 d1
  Surgery:
  Scheduled 6-8 weeks after the completion of CRT Adjuvant Chemotherapy: depends on patients pathological review.
  Interventions: Radiation: Pelvic Radiation; Drug: Capecitabine; Drug: Irinotecan; Other: Placebo

INTERVENTIONS:
Drug: Dendrobium Huoshanense Granules — 3g tid per day for 5weeks
  Arms: CRT with Dendrobium Huoshanense
Radiation: Pelvic Radiation — 50Gy/25Fx
Drug: Capecitabine — 625mg/m2 bid Monday-Friday per week
Drug: Irinotecan — 80mg/m2 (UGT1A1*28 6/6) or 65mg/m2 (UGT1A1*28 6/7)
Other: Placebo — 3g tid per day for 5weeks
  Arms: CRT with Placebo

SUMMARY:
The study evaluates the addition of Chinese Herbal Compound Dendrobium Huoshanense Granules to capecitabine and irinotecan in neoadjuvant chemoradiation(CRT) in locally advanced rectal cancer. Half of participants will receive CRT with Dendrobium Huoshanense Granules, while the others will receive CRT with placebo. We will evaluate whether Dendrobium Huoshanense Granules can enhance the immune function and alleviate symptoms caused by the tumor and CRT .

ELIGIBILITY:
Inclusion Criteria:

* pathological confirmed rectum adenocarcinoma
* clinical stage T3-4 and/or N+
* the distance from anal verge less than 10 cm
* without distance metastases
* performance status score: 0~1
* UGT1A1*28 6/6 or 6/7
* without previous anti-cancer therapy
* able to follow the protocol during the study period
* sign the inform consent

Exclusion Criteria:

* Pregnant or breastfeeding women
* Those with other history of malignant disease in the past 5 years, except for cured skin cancer and cervical carcinoma in situ
* If there is an uncontrolled history of epilepsy, central nervous system disease or mental disorder, the investigator may determine that the clinical severity may hinder the signing of informed consent or affect the patient's oral medication compliance.
* Clinically severe (ie, active) heart disease, such as symptomatic coronary heart disease, New York Heart Association (NYHA) class II or more severe congestive heart failure or severe arrhythmia requiring medication intervention (see appendix 12), or a history of myocardial infarction in the last 12 months
* Organ transplantation requires immunosuppressive therapy
* Severe uncontrolled recurrent infections, or other serious uncontrolled concomitant diseases
* Subject blood routine and biochemical indicators do not meet the following criteria: hemoglobin ≥ 90g / L; absolute neutrophil count (ANC) ≥ 1.5 × 109 / L; Alanine transaminase (ALT), aspartate aminotransferase (AST) ≤ 2.5 times the upper limit of normal; alkaline phosphatase (ALP) ≤2.5 times the normal upper limit; serum total bilirubin <1.5 times the normal upper limit; serum creatinine <1 times the normal upper limit; serum albumin ≥ 30g / L
* Anyone who is allergic to any research medication
* DPD deficiency
* UGT1A1*28 7/7

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
the morbidity of hematological adverse events and diarrhea as assessed by CTCAE v4.0 | twice weekly during the neoadjuvant chemotherapy (5 weeks)

SECONDARY OUTCOMES:
Impact of participants' quality of life during treatment as assessed by EQ-5D questionnaire | once weekly during the neoadjuvant chemotherapy (5 weeks)
Impact of participants' quality of life during treatment as assessed by EORTC-QLQ-C30 questionnaire | once weekly during the neoadjuvant chemotherapy (5 weeks)
ORR(objective response rate) includes CR(complete rate) and PR(partial rate) | Surgery scheduled 6-8 weeks after the end of chemoradiation
Number of the concurrent chemotherapy cycles that patients can receive during radiotherapy | once weekly during neoadjuvant chemoradiation(5 weeks,each cycle is one week)

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Zhang, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China